CLINICAL TRIAL: NCT04963400
Title: Impact of Hospitalization on High-sensitivity Cardiac Troponin T Concentrations Depending on Disease Severity (Inpatient Troponin T)
Brief Title: Impact of Hospitalization on High-sensitivity Cardiac Troponin T Concentrations Depending on Disease Severity
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Rolf Wachter, Professor MD, University of Leipzig
Other Study IDs: RL_2021_1
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Non-cardiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with low disease severity: Hospitalized patients without a diagnosed or suspected cardiac disease and with an acute medical condition of low severity (e.g. patients with retinal detachment)
  Interventions: Diagnostic Test: Analysis of hs-cTnT serum concentration at hospitalization; Diagnostic Test: Analysis of hs-cTnT serum concentration after discharge
- Patients with medium disease severity: Hospitalized patients without a diagnosed or suspected cardiac disease and with an acute medical condition of medium severity (e.g. patients with an uncomplicated acute pancreatitis oder an acute exacerbation of a chronic inflammatory bowel disease)
  Interventions: Diagnostic Test: Analysis of hs-cTnT serum concentration at hospitalization; Diagnostic Test: Analysis of hs-cTnT serum concentration after discharge
- Patients with high disease severity: Hospitalized patients without a diagnosed or suspected cardiac disease and with an acute medical condition of high severity (e.g. patients with a proximal femoral fracture)
  Interventions: Diagnostic Test: Analysis of hs-cTnT serum concentration at hospitalization; Diagnostic Test: Analysis of hs-cTnT serum concentration after discharge

INTERVENTIONS:
Diagnostic Test: Analysis of hs-cTnT serum concentration at hospitalization — Analysis of the hs-cTnT serum concentration in the blood drawn at the day of hospitalization
Diagnostic Test: Analysis of hs-cTnT serum concentration after discharge — Analysis of the hs-cTnT serum concentration in the blood drawn after discharge (60 days after hospitalization)

SUMMARY:
We aim to examine, whether hospitalization is associated with higher high-sensitivity cardiac troponin T (hs-cTnT) serum concentrations in patients without a cardiac disease.

DETAILED DESCRIPTION:
High-sensitivity cardiac troponin T (hs-cTnT) values will be obtained in hospitalized patients a) without a diagnosed or suspected cardiac disease, and b) with an acute medical condition that is not commonly associated with an increase of hs-cTnT concentrations. As a reference, a second sampling of blood for an analysis of the hs-cTnT serum concentration will be obtained in the same patients after discharge (60 days after hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* hospitalization due to a non-cardiac disease
* age ≥ 50 years

Exclusion Criteria:

* diagnosed or suspected cardiac disease
* acute medical conditions commonly associated with a myocardial injury (e.g. circulatory shock, sepsis, pulmonary embolism, cerebral infarction, acute renal failure)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 312 patients with an acute, non-cardiac medical condition of low, medium or high severity (104 patients per group)
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Difference of the hs-cTnT concentration at hospitalization and after discharge | 60 days

SECONDARY OUTCOMES:
Difference of the hs-cTnT concentration at hospitalization and after discharge in acute medical conditions of low severity | 60 days
Difference of the hs-cTnT concentration at hospitalization and after discharge in acute medical conditions of medium severity | 60 days
Difference of the hs-cTnT concentration at hospitalization and after discharge in acute medical conditions of high severity | 60 days
Prediction of 1-year-mortality by hs-cTnT concentration | 1 year
Prediction of 1-year-hospitalization rate due to a cardiovascular disease by hs-cTnT concentration | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig Medical Center, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable scientific request